CLINICAL TRIAL: NCT02238210
Title: A Phase IV Safety Trial in Pediatric Patients (Ages 2-5) With Rhinorrhea Associated With a Common Cold or Allergy
Brief Title: Safety Trial of Atrovent® in Pediatric Patients With Rhinorrhea Associated With a Common Cold or Allergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 244.2503
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Cold
MeSH Terms: conditions — Common Cold | interventions — Ipratropium

ARMS (2):
- Atrovent® - common cold group (Experimental): Treatment duration for common cold group - three time daily for 4 days
  Interventions: Drug: Atrovent®
- Experimental: Atrovent® - allergy group (Experimental): Treatment duration for allergy group - three time daily for 14 days
  Interventions: Drug: Atrovent®

INTERVENTIONS:
Drug: Atrovent®

SUMMARY:
Study to determine the safety of Atrovent Nasal Spray 0.06% in pediatric patients (ages 2-5 years) with symptoms of rhinorrhea associated with a naturally occurring common cold or from symptoms of rhinorrhea associated with allergies

ELIGIBILITY:
Inclusion Criteria for patients with common cold

* Male or female at least 2 but not older than 5 years of age at screening
* Have a diagnosis of a common cold defined as presence of acute onset of rhinorrhea (within 48 hours of screening visit) and at least 1 of the following:

  * Presence of swollen nasal membranes characteristic of a common cold on examination at screening
  * Presence of fever up to 102°F (oral or equivalent) within 48 hours of visit (may be taken at home/away from the clinic) or at time of screening
* Capability of parent/legal guardian to read and understand the informed consent, record trial diary information, administer trial drug and read and understand trial assessment questionnaire

Inclusion Criteria for patients with allergies

* Male or female at least 2 but not older than 5 year of age
* Have a diagnosis of seasonal or perennial allergic rhinitis defined as having both of the following:

  * Positive skin or Radioallergosorbent test (RAST) test to a relevant allergen within 12 months of screening or at the screening visit. For the purpose of this trial a positive skin test is defined as wheal diameter that is at least 3 mm greater than the negative control
  * Positive prior history for atopy with nasal symptoms associated with expose to allergens
* Symptoms associated with rhinorrhea for at least 48 hours prior to the screening visit
* Capability of parent/legal guardian to read and understand the informed consent, record trial diary information, administer trial drug and read and understand trial assessment questionnaire

General Exclusion Criteria for both common cold and allergy

* Significant cardiovascular, renal, hepatic, endocrine, metabolic, neurologic or other systemic disease. A significant disease was defined as one which, in the opinion of the Investigator, either put the patient at risk because of participation in the trial or influenced the results of the trial or the patient's ability to participate in the trial
* Presence of rales or rhonchi suggestive of a lower respiratory tract infection
* An oral (or equivalent) temperature higher than 102°F
* Presence of otitis media
* Be initiating or advancing immunotherapy regimen during the course of this trial. Patients receiving a maintenance dose of immunotherapy are eligible
* Known intolerance to anticholinergics of hypersensitivity to benzalkonium chloride
* Excluded medications prior to Visit 1 and during the trial included:

  1. 24 hours before

     * Over-the-counter decongestants or nasal/ocular cromolyn
  2. 3 days before:

     * Anticholinergics
     * Over-the-counter antihistamines
     * sympathomimetic decongestants
  3. 5 days before:

     * Fexofenadine
     * Loratadine
  4. 7 days before:

     * Cetirizine
     * antihistamines such as Atarax® or doxepin hydrochloride
     * Antidepressants
  5. 14 days before:

     * Intranasal steroids
  6. 28 days before:

     * Steroids (oral and injectable)
     * Leukotriene modifiers (e.g. Accolate®, Singulair®)
     * Other investigational drugs
* Participation in any trial with an investigational drug within 30 days of the screening visit
* Nasal obstruction greater than 50% that would prevent deposition of trial drug
* The parent/legal guardian has a disability or lives in a geographical location that could impair compliance with the protocol or visits to the trial center

Exclusion criteria for patients with a common cold

* History or perennial allergic rhinitis or seasonal allergic rhinitis (SAR) with allergen in season
* Positive Streptococcus test

Exclusion criteria for patients with allergies

* Patients with active infectious rhinitis (common cold) as determined by history and physical
* Patients with upper or lower respiratory infection at screening

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2002-12; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Patient's parent/legal guardian global assessment - common cold group | Day 4
Number of patients with adverse events | up to 21 days
Patient's parent/legal guardian global assessment - allergy group | Day 14

SECONDARY OUTCOMES:
Patient's parent/legal guardian daily assessment of rhinorrhea (runny nose) rated on 5-point scale - common cold group | Day 4
  daily assessment by e-diary
Patient's parent/legal guardian daily assessment of nasal congestion (stuffy nose) rated on 5-point scale - common cold group | Day 4
  daily assessment by e-diary
Patient's parent/legal guardian daily assessment of sneezing rated on 5-point scale - common cold group | Day 4
  daily assessment by e-diary
Number of patients with clinically findings in nasal and otoscopic examination - common cold group | up to day 4
Patient's parent/legal guardian daily assessment of rhinorrhea (runny nose) rated on 5-point scale - allergy group | Day 14
  daily assessment by e-diary
Patient's parent/legal guardian daily assessment of nasal congestion (stuffy nose) rated on 5-point scale - allergy group | Day 14
  daily assessment by e-diary
Patient's parent/legal guardian daily assessment of sneezing rated on 5-point scale - allergy group | Day 14
  daily assessment by e-diary
Number of patients with clinically findings in nasal and otoscopic examination - allergy group | up to day 14